CLINICAL TRIAL: NCT00466947
Title: COMPAS: A Phase III Study to Demonstrate Efficacy of GSK Biologicals' 10-valent Pneumococcal Vaccine (GSK1024850A) Against Community Acquired Pneumonia and Acute Otitis Media
Brief Title: COMPAS (Clinical Otitis Media & Pneumonia Study): Pneumonia & Acute Otitis Media (AOM ) Efficacy Study of the Pneumococcal Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 109563; 2011-002076-16 (EudraCT Number)
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Results first posted 2013-09-04 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Infections, Streptococcal
Keywords: Otitis media; Pneumonia; Community acquired pneumonia (CAP); Pneumococcal disease; Booster vaccination; Immunogenicity; Pneumococcal vaccine; Safety; Efficacy; Carriage
MeSH Terms: conditions — Streptococcal Infections; Otitis Media; Pneumonia; Community-Acquired Pneumonia; Pneumococcal Infections | interventions — Hepatitis A Vaccines; Engerix-B; Hepatitis B Vaccines; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

STUDY DESIGN:
Who Masked: Care Provider, Investigator

ARMS (2):
- Synflorix Group (Experimental): Subjects received 3 primary doses of Synflorix at 2, 4 and 6 months of age co-administered with Infanrix-hexa and booster dose of Synflorix at 15-18 months of age co-administered with Infanrix-IPV/Hib. All vaccines were administered intramuscularly in the right (Synflorix) or the left (Infanrix-hexa, Infanrix-IPV/Hib) thigh (primary dose) or deltoid (booster dose).
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A; Biological: Havrix; Biological: Infanrix hexa; Biological: GSK Biologicals' DTPa-IPV/Hib vaccine
- Control Group (Active Comparator): Subjects received 3 doses of Engerix at 2, 4 and 6 months of age co-administered with Infanrix-IPV/Hib and 1 dose of Havrix co-administered with Infanrix-IPV/Hib at 15-18 months of age. All vaccines were administered in the right (Engerix, Havrix) or the left (Infanrix-IPV/Hib) thigh.
  Interventions: Biological: Havrix; Biological: Engerix-B; Biological: GSK Biologicals' DTPa-IPV/Hib vaccine

INTERVENTIONS:
Biological: Pneumococcal conjugate vaccine GSK1024850A — Intramuscular injection, 4 doses
  Arms: Synflorix Group
Biological: Havrix — Intramuscular injection, 2 doses in Synflorix group and 3 doses in Control group
  Other Names: Hepatitis A vaccine
Biological: Engerix-B — Intramuscular injection, 3 doses
  Other Names: Hepatitis B vaccine
  Arms: Control Group
Biological: Infanrix hexa — Intramuscular injection,3 doses
  Other Names: DTPa-HBV-IPV/Hib
  Arms: Synflorix Group
Biological: GSK Biologicals' DTPa-IPV/Hib vaccine — Intramuscular injection, 1 dose in Synflorix group and 4 doses in Control group

SUMMARY:
This is a study in a large number of healthy children less than 3 years old to measure the efficacy of GlaxoSmithKline (GSK) Biologicals' 10-valent pneumococcal conjugate candidate vaccine (Synflorix vaccine, or GSK1024850A) to prevent cases of pneumonia (lung infection) likely caused by bacteria (Streptococcus pneumoniae and Haemophilus influenzae) or cases of otitis media (ear infection) in children under 3 years old.

DETAILED DESCRIPTION:
The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007. The following vaccines will be offered by the sponsor:

* Two doses of hepatitis A vaccine will be offered to all subjects to comply with national recommendations.
* NeisVac-C vaccine against Neisseria meningitis group C will be offered to all subjects in Argentina at 12 months of age.
* Varicella vaccine will be offered to all subjects in Colombia and Panama at 12 months of age.
* Two doses of Rotarix vaccine will be offered to all subjects in Colombia within the first six months of life.

In addition, all subjects will receive a dose of Hepatitis B vaccine at birth according to national recommendations and a dose of measles, mumps and rubella (MMR) vaccine at 12 to 15 months of age according to local Extended Program of Immunization (EPI) .

These vaccines will not be provided by the sponsor. The protocol posting has been updated according to the amendment of the protocol dated 25 Nov 2008. The protocol posting has been updated according to the amendment of the protocol dated 14 December 2009. The protocol posting has been updated according to the amendment of the protocol dated 09 September 2010.

ELIGIBILITY:
Inclusion Criteria:

* A male or female between, and including, 6 and 16 weeks of age at the time of the first vaccination. Pre-term born infants can be included in the study starting from 8 weeks of chronological age at the time of first vaccination and up to 16 weeks of chronological age
* Subjects should be living in the area covered by the surveillance system for community acquired pneumonia (CAP), invasive disease and acute otitis media (AOM) •Written informed consent obtained from the parent or guardian of the subject.
* Free of any known or suspected health problems (as established by medical history and clinical examination before entering into the study), that would contraindicate the initiation of routine immunizations outside a clinical trial context.
* Subjects for whom the investigator believes that their parents/guardians can and will comply with the requirements of the protocol

Exclusion Criteria:

* Use of any investigational or non-registered drug or planned use during the study period.
* Use or planned use of any investigational or non-registered vaccine other than the study vaccine(s).
* Previous vaccination against diphtheria, tetanus, pertussis, Haemophilus influenzae type b, hepatitis A and/or Streptococcus. pneumoniae . Locally recommended EPI vaccines to be given at birth are allowed, but should be administered at least one month before the first dose of the study vaccine .Other locally recommended vaccines are always allowed, even if concomitantly administered with the study vaccines. •Previous or planned vaccination with a registered pneumococcal vaccine such as Prevnar is not allowed. If Prevnar immunization needs to be initiated, due to the presence of a high risk disease for pneumococcal infections for which the Prevnar vaccine is made locally available, the subject can not be enrolled in the study and should be referred to the specific Prevnar immunization program.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment
* For Colombia: infants with low birth weight ( less than (<) 2.500 grams)

Ages: 6 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23802 (Actual)
Dates: Start 2007-06-28 (Actual); Primary Completion 2010-08-31 (Actual); Study Completion 2011-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (18):
- Argentina (16):
  - GSK Investigational Site, Godoy Cruz, Mendoza Province
  - GSK Investigational Site, Las Heras, Mendoza Province
  - GSK Investigational Site, Luján de Cuyo, Mendoza Province
  - GSK Investigational Site, Villa Nueva, Mendoza Province
  - GSK Investigational Site, Villanueva, Mendoza Province
  - GSK Investigational Site, Albardón, San Juan Province
  - GSK Investigational Site, Caucete, San Juan Province
  - GSK Investigational Site, Fernández, Santiago del Estero Province
  - GSK Investigational Site, La Banda, Santiago del Estero Province
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, La Banda
  - GSK Investigational Site, Maipú
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Juan
  - GSK Investigational Site, San Martín
  - GSK Investigational Site, Santiago del Estero
- GSK Investigational Site, Cali, Colombia
- GSK Investigational Site, Panama City, Panama

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Silfverdal SA, Coremans V, Francois N, Borys D, Cleerbout J. Safety profile of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV). Expert Rev Vaccines. 2017 Feb;16(2):109-121. doi: 10.1586/14760584.2016.1164044. Epub 2016 Sep 30. PMID 26954689
- [Background] Saez-Llorens X, Rowley S, Wong D, Rodriguez M, Calvo A, Troitino M, Salas A, Vega V, Castrejon MM, Lommel P, Pascal TG, Hausdorff WP, Borys D, Ruiz-Guinazu J, Ortega-Barria E, Yarzabal JP, Schuerman L. Efficacy of 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine against acute otitis media and nasopharyngeal carriage in Panamanian children - A randomized controlled trial. Hum Vaccin Immunother. 2017 Jun 3;13(6):1-16. doi: 10.1080/21645515.2017.1287640. Epub 2017 Feb 25. PMID 28368738
- [Background] Tregnaghi MW, Saez-Llorens X, Lopez P, Abate H, Smith E, Posleman A, Calvo A, Wong D, Cortes-Barbosa C, Ceballos A, Tregnaghi M, Sierra A, Rodriguez M, Troitino M, Carabajal C, Falaschi A, Leandro A, Castrejon MM, Lepetic A, Lommel P, Hausdorff WP, Borys D, Ruiz Guinazu J, Ortega-Barria E, Yarzabal JP, Schuerman L; COMPAS Group. Efficacy of pneumococcal nontypable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) in young Latin American children: A double-blind randomized controlled trial. PLoS Med. 2014 Jun 3;11(6):e1001657. doi: 10.1371/journal.pmed.1001657. eCollection 2014 Jun. PMID 24892763
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 109563 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109563 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109563 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109563 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109563 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109563 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Analysis on the primary outcome was performed when at least 535 first bacterial CAP episodes were reported from 2 weeks after vaccine Dose 3 (31 August 2010) with 23738 subjects (11875 and 11863 in Synflorix and Control groups) and analysis at study end was performed on 23597 subjects.
Groups:
- Control Group: Subjects received 3 doses of Engerix at 2,4 and 6 months of age co-administered with Infanrix-IPV/Hib and 1 dose of Havrix co-administered with Infanrix-IPV/Hib at 15-18 months of age. All vaccine were administered in the right (Engerix, Havrix) or the left (Infanrix-IPV/Hib) thigh.
Period: Primary Outcome Analysis Period
Arm/Group | Synflorix Group | Control Group
Started | 11875 | 11863
Ongoing | 11875 | 11863
Completed | 0 (No data on study completion and withdrawal were available at first analysis as the study was ongoing) | 0 (No data on study completion and withdrawal were available at first analysis as the study was ongoing)
Not Completed | 11875 | 11863
Not completed — Other: study still ongoing | 11875 | 11863
Period: Study End Analysis Period
Arm/Group | Synflorix Group | Control Group
Started | 11798 | 11799
Completed | 9302 | 9265
Not Completed | 2496 | 2534
Not completed — Adverse Event | 35 | 43
Not completed — Lost to Follow-up | 1137 | 1167
Not completed — Physician Decision | 29 | 29
Not completed — Protocol Violation | 9 | 17
Not completed — Withdrawal by Subject | 1264 | 1267
Not completed — Other - Forbidden vaccination | 21 | 10
Not completed — Other - Subject without a legal guardian | 1 | 0
Not completed — Other - Unconformity in team's treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix Group | Control Group | Total
Number analyzed (Participants) | 11798 | 11799 | 23597
Age, Continuous [Mean (Standard Deviation); unit: Weeks] — Baseline measures presented below correspond to those of the subjects whose data were exploited towards analysis of results at the end of the study
  Weeks | 9.2 (1.93) | 9.2 (1.92) | 9.2 (1.92)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline measures presented below correspond to those of the subjects whose data were exploited towards analysis of results at the end of the study
  Participants
    Female | 5796 | 5767 | 11563
    Male | 6002 | 6032 | 12034
Region of Enrollment [Number; unit: Subjects] — Baseline measures presented below correspond to those of the subjects whose data were exploited towards analysis of results at the end of the study
  Subjects
    Argentina | 6990 | 6991 | 13981
    Columbia | 1206 | 1196 | 2402
    Panama | 3602 | 3612 | 7214

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a First Episode Reported of Bacterial Community Acquired Pneumoniae (B-CAP)
Description: A B-CAP episode was defined as a radiologically confirmed community acquired pneumoniae (CAP) episode with either alveolar consolidation/pleural effusion on the chest X-ray (CXR) or with non-alveolar infiltrates but with C reactive protein (CRP) higher than or equal to (>=) 40 milligrams per liter (mg/L). The results are presented for data lock point for the primary outcome analysis (31 August 2010), which was performed, as per protocol, when at least 535 first B-CAP episodes were reported from 2 weeks after the third vaccination dose. After analysis on primary outcome was performed, re-monitoring activities revealed Informed Consent Form issues for some subjects. Therefore, a sensitivity analysis excluding 144 subjects was performed. This analysis confirmed the validity of the results for primary outcome.
Time Frame: Any time from 2 weeks after Dose 3 up to 31 August 2010
Population: Analysis was performed on the Interim ATP cohort for efficacy which included all evaluable vaccinated subjects who had received the 3-dose primary vaccination course, with available contact and efficacy data beyond Day 14 post study vaccine Dose 3, and whose parents/guardians consented to the use of the subject's data as of 31 August 2010.
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 10295 | 10201
Subjects | 240 | 304

2. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Throughout the study (Month 0 to Month 22-25)
Population: The analysis was performed on all vaccinated subjects whose data were exploited towards analysis of results at the end of the study.
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 11798 | 11799
Subjects | 2534 | 2668

3. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Event (AE), in the Panama Subset
Description: An unsolicited AE is any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. The Panama Subset included all subjects from Panama.
Time Frame: Throughout the study (Month 0 to Month 22-25)
Population: The analysis was performed on all vaccinated subjects included in the Panama subset.
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 3602 | 3612
Subjects | 3530 | 3518

4. Secondary Outcome: Number of Subjects With Solicited Local Symptoms Post Primary Vaccination in the Immunogenicity and Tolerability Subset
Description: Assessed symptoms were redness, swelling and pain. The Immunogenicity and Tolerability Subset included 500 subjects coming from Argentina and Panama respectively. This outcome measure concerns solely subjects from the Synflorix Group.
Time Frame: Within the 4-days (Days 0-3) follow-up period across the 3 doses of the primary study vaccine administration
Population: The analysis was performed on all vaccinated subjects included in the Immunogenicity and Tolerability subset for the primary vaccination course.
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group
Number analyzed (Participants) | 368
Subjects
  Pain after vaccination with Synflorix | 275
  Pain after vaccination with Infanrix Hexa | 270
  Redness after vaccination with Synflorix | 182
  Redness after vaccination with Infanrix Hexa | 171
  Swelling after vaccination with Synflorix | 141
  Swelling after vaccination with Infanrix Hexa | 143

5. Secondary Outcome: Number of Subjects With Solicited Local Symptoms Post Booster Vaccination in the Immunogenicity and Tolerability Subset
Description: as for outcome 4
Time Frame: Within the 4-days (Days 0-3) follow-up period following the booster vaccine administration
Population: The analysis was performed on all vaccinated subjects included in the Immunogenicity and Tolerability subset for the booster vaccination.
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group
Number analyzed (Participants) | 317
Subjects
  Pain after vaccination with Synflorix | 129
  Pain after vaccination with Infanrix-IPV/Hib | 131
  Redness after vaccination with Synflorix | 104
  Redness after vaccination with Infanrix-IPV/Hib | 98
  Swelling after vaccination with Synflorix | 74
  Swelling after vaccination with Infanrix-IPV/Hib | 69

6. Secondary Outcome: Number of Subjects With Solicited Local Symptoms Post Primary Vaccination in the Immunogenicity and Tolerability Subset
Description: Assessed symptoms were redness, swelling and pain. The Immunogenicity and Tolerability Subset included 500 subjects coming from Argentina and Panama respectively. This outcome measure concerns solely subjects from the Control Group.
Time Frame: Within the 4-days (Days 0-3) follow-up period across the 3 doses of the primary study vaccine administration
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Control Group
Number analyzed (Participants) | 357
Subjects
  Pain after vaccination with Infanrix-IPV/Hib | 169
  Pain after vaccination with Engerix | 165
  Redness after vaccination with Infanrix-IPV/Hib | 118
  Redness after vaccination with Engerix | 109
  Swelling after vaccination with Infanrix-IPV/Hib | 98
  Swelling after vaccination with Engerix | 91

7. Secondary Outcome: Number of Subjects With Solicited Local Symptoms Post Booster Vaccination in the Immunogenicity and Tolerability Subset, for the Control Group
Description: Assessed symptoms were redness, swelling and pain. The Immunogenicity and Safety Tolerability Subset included 500 subjects coming from Argentina and Panama respectively. This outcome measure concerns solely subjects from the Control Group.
Time Frame: Within the 4-days (Days 0-3) follow-up period following the booster vaccine administration.
Population: as for outcome 5
Measure: Number; unit: Subjects
Arm/Group | Control Group
Number analyzed (Participants) | 303
Subjects
  Pain after vaccination with Infanrix-IPV/Hib | 81
  Pain after vaccination with Havrix | 89
  Redness after vaccination with Infanrix-IPV/Hib | 81
  Redness after vaccination with Havrix | 73
  Swelling after vaccination with Infanrix-IPV/Hib | 70
  Swelling after vaccination with Havrix | 55

8. Secondary Outcome: Number of Subjects With Solicited General Symptoms Post Primary Vaccination in the Immunogenicity and Tolerability Subset
Description: Assessed symptoms were fever (defined as rectal temperature equal or higher than [>=] 38 degrees Celsius [°C]). irritability/fussiness, drowsiness, and loss of appetite. The Immunogenicity and Tolerability Subset included 500 subjects coming from Argentina and Panama respectively.
Time Frame: Within the 4-days (Days 0-3) follow-up period across the 3 doses of the primary study vaccine administration
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 368 | 357
Subjects
  Drowsiness | 236 | 168
  Fever (rectal temperature >= 38°C) | 247 | 125
  Irritability | 289 | 206
  Loss of appetite | 133 | 80

9. Secondary Outcome: Number of Subjects With Solicited General Symptoms Post Booster Vaccination in the Immunogenicity and Tolerability Subset
Description: as for outcome 8
Time Frame: Within the 4-days (Days 0-3) follow-up period following the booster vaccine administration
Population: as for outcome 5
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 317 | 303
Subjects
  Drowsiness | 74 | 65
  Fever (rectal temperature >= 38°C) | 93 | 73
  Irritability | 121 | 95
  Loss of appetite | 51 | 46

10. Secondary Outcome: Number of Subjects With a First Episode Reported of Clinically Confirmed Acute Otitis Media (AOM) (C-AOM), in the Panama Subset
Description: The Panama Subset contained all subjects enrolled in Panama.
Time Frame: Any time from 2 weeks after Dose 3 to study end at Month 22-25
Population: Analysis was performed on the Final ATP cohort for efficacy which included all evaluable vaccinated subjects who had received the 3-dose primary vaccination course, with available contact and efficacy data beyond Day 14 post study vaccine Dose 3, and whose parents/guardians consented to the use of the subject's data as of study end.
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 3010 | 2979
Subjects | 204 | 239

11. Secondary Outcome: Number of Subjects With a First Episode Reported of Community Acquired Pneumoniae (CAP) With Alveolar Consolidation or Pleural Effusion on the Chest X-ray (CXR) (C-CAP)
Description: CXR alveolar consolidation was defined as CXR with a dense, often homogeneous, confluent alveolar infiltrate that could encompass an entire lobe or segment, or a fluffy, mass-like, cloud-like density that erased heart and diaphragm borders (silhouette sign) and that often contained air bronchograms. CXR pleural effusion was defined as a fluid collecting in the pleural space around the lung, seen radiologically as a dense rim (the same density as the chest-wall muscles) interposed between the lung and the ribs.
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 10211 | 10140
Subjects | 181 | 231

12. Secondary Outcome: Number of Subjects With a First Episode Reported of Bacteriologically Confirmed Acute Otitis Media (AOM) (B-AOM) Due to Any Bacterial Pathogen, in the Panama Subset
Description: The Panama Subset contained all subjects enrolled in Panama.
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 3010 | 2979
Subjects | 32 | 45

13. Secondary Outcome: Number of Subjects With a First Episode Reported of Bacteriologically Confirmed Acute Otitis Media (AOM) (B-AOM) Due to Streptococcus Pneumoniae (S. pn.) Vaccine Serotypes, in the Panama Subset
Description: The 10 pneumococcal S. pneumoniae vaccine serotypes assessed for this outcome measure were the serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. The Panama Subset contained all subjects enrolled in Panama.
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 3010 | 2979
Subjects | 6 | 18

14. Secondary Outcome: Number of Subjects With a First Episode Reported of Bacteriologically Confirmed Acute Otitis Media (AOM) (B-AOM) Due to Streptococcus Pneumoniae (S. pn.) Cross-reactive Serotypes, in the Panama Subset.
Description: The S. pn. cross-reactive serotypes assessed for this outcome measure were the serotypes 6A, 18B, 19A and 23A. The Panama Subset contained all subjects enrolled in Panama.
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 3010 | 2979
Subjects | 3 | 4

15. Secondary Outcome: Number of Subjects With a First Episode Reported of Bacteriologically Confirmed Acute Otitis Media (AOM) (B-AOM) Due to Other Pneumococcal Serotypes, in the Panama Subset.
Description: Other pneumococcal serotypes were defined for this outcome measures as non-Streptococcus pneumoniae vaccine and cross-reactive serotypes. The Panama Subset contained all subjects enrolled in Panama.
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 3010 | 2979
Subjects | 3 | 4

16. Secondary Outcome: Number of Subjects With a First Episode Reported of Bacteriologically Confirmed Acute Otitis Media (AOM) (B-AOM) Due to Haemophilus Influenzae (H. Influenzae), in the Panama Subset
Description: The Panama Subset contained all subjects enrolled in Panama.
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 3010 | 2979
Subjects | 12 | 14

17. Secondary Outcome: Number of Subjects With a First Episode Reported of Bacteriologically Confirmed Acute Otitis Media (AOM) (B-AOM) Due to Non-typeable Haemophilus Influenzae (H. Influenzae), in the Panama Subset
Description: The Panama Subset contained all subjects enrolled in Panama
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 3010 | 2979
Subjects | 12 | 14

18. Secondary Outcome: Number of Subjects With a First Episode Reported of Bacteriologically Confirmed Acute Otitis Media (AOM) (B-AOM) Due to Other AOM Pathogens, in the Panama Subset
Description: Other pathogens assessed included among others Moraxella catarrhalis, Group A streptococci, and Staphyloccus aureus. The Panama Subset contained all subjects enrolled in Panama.
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 3010 | 2979
Subjects | 8 | 7

19. Secondary Outcome: Number of Subjects With a First Episode Reported of Community Acquired Pneumoniae (CAP) With Alveolar Consolidation or Pleural Effusion on the Chest X-ray (CXR) (C-CAP) With Positive Respiratory Viral Test (RVT)
Description: A CXR with consolidation was defined as a CXR with a dense, often homogeneous, confluent alveolar infiltrate that could encompass an entire lobe or segment, or a fluffy, mass-like, cloud-like density that erased heart and diaphragm borders (silhouette sign) and that often contained air bronchograms. Pleural effusion was defined as a fluid collecting in the pleural space around the lung, seen radiologically as a dense rim (the same density as the chest-wall muscles) interposed between the lung and the ribs.
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 10211 | 10140
Subjects | 21 | 25

20. Secondary Outcome: Number of Subjects With a First Episode Reported of Community Acquired Pneumoniae (CAP) With Any Abnormal CXR With Positive Respiratory Viral Test (RVT)
Description: An "abnormal CXR" was defined as a CXR with either consolidation, pleural effusion and/or abnormal pulmonary alveolar or non-alveolar infiltrates on the digital CXR image. CXR with consolidation was defined as a CXR with a dense, often homogeneous, confluent alveolar infiltrate that could encompass an entire lobe or segment, or a fluffy, mass-like, cloud-like density that erased heart and diaphragm borders (silhouette sign) and that often contained air bronchograms. Pleural effusion was defined as a fluid collecting in the pleural space around the lung, seen radiologically as a dense rim (the same density as the chest-wall muscles) interposed between the lung and the ribs.
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 10211 | 10140
Subjects | 104 | 112

21. Secondary Outcome: Number of Subjects With a First Episode Reported of Bacterial Community Acquired Pneumoniae (B-CAP) With Positive Respiratory Viral Test (RVT).
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 10211 | 10140
Subjects | 35 | 39

22. Secondary Outcome: Number of Subjects With a First Episode Reported of Suspected Community Acquired Pneumoniae (CAP) (S-CAP)
Description: An episode of S-CAP involved either any subject who was referred to have a chest X-ray (CXR) performed as part of the clinical assessment of a febrile syndrome or an acute respiratory infection (ARI), or a hospitalized child who had a CXR performed within 2 days prior to, or within the first 3 days after hospital admission, as part of the clinical assessment of a febrile syndrome or an ARI.
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 10211 | 10140
Subjects | 2108 | 2237

23. Secondary Outcome: Number of Subjects With a First Episode Reported of Community Acquired Pneumoniae (CAP) With Any Abnormal Chest X-ray (CXR)
Description: as for outcome 20
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 10211 | 10140
Subjects | 681 | 764

24. Secondary Outcome: Number of Subjects With a First Episode Reported of Suspected Community Acquired Pneumoniae (CAP) (S-CAP) With C Reactive Protein (CRP) >= Cut-off, Regardless of Chest X-ray (CXR) Reading
Description: A case of S-CAP involved either any subject who was referred to have a CXR performed as part of the clinical assessment of a febrile syndrome or an acute respiratory infection (ARI), or a hospitalized child who had a CXR performed within 2 days prior to, or within the first 3 days after hospital admission, as part of the clinical assessment of a febrile syndrome or an ARI. CRP cut-off values applied for this outcome measure were 40 milligrams per liter (mg/L), 80 mg/L, and 120 mg/L.
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 10211 | 10140
Subjects
  S-CAP with CRP >= 40 mg/L regardless of CXR exam | 425 | 499
  S-CAP with CRP >= 80 mg/L regardless of CXR exam | 175 | 237
  S-CAP with CRP >= 120 mg/L regardless of CXR exam | 85 | 119

25. Secondary Outcome: Number of Subjects With a First Episode Reported of CAP With Either Alveolar Consolidation/Pleural Effusion on Chest X-ray (CXR) (C-CAP) or With Non-alveolar Infiltrates (NAI-CAP) But With C Reactive Protein (CRP) >= Cut-off.
Description: CRP cut-off values applied for this outcome measure were 80 milligrams per liter (mg/L), and 120 mg/L.
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 10211 | 10140
Subjects
  C-CAP or NAI-CAP with CRP >= 80 mg/L | 208 | 256
  C-CAP or NAI-CAP with CRP >= 120 mg/L | 191 | 240

26. Secondary Outcome: Number of Subjects With a First Episode Reported of Vaccine-type Invasive Pneumococcal Disease (VT-IPD).
Description: A VT-IPD was defined as a bacteriologically culture confirmed invasive pneumococcal disease case caused by any of the 10 pneumococcal Streptococcus pneumoniae vaccine serotypes. The 10 pneumococcal S. pneumoniae vaccine serotypes assessed for this outcome measure were the serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 10211 | 10140
Subjects | 0 | 16

27. Secondary Outcome: Number of Subjects With a First Episode Reported of a Bacteriologically Confirmed Invasive Pneumococcal Disease (Bact.-Conf. ID).
Description: A Bact.-conf. ID was defined as a bacteriologically culture confirmed invasive pneumococcal disease (ID) cases due to any of the 10 Streptococcus pneumoniae vaccine serotypes as identified through positive culture. The 10 pneumococcal S. pneumoniae vaccine serotypes assessed for this outcome measure were the serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 10211 | 10140
Subjects | 6 | 17

28. Secondary Outcome: Number of Subjects With a First Episode Reported of Pneumococcal Invasive Disease (Pneumococcal ID)
Description: A Pneumococcal ID was defined as a bacteriologically culture confirmed invasive pneumococcal disease (ID) cases due to any of the 10 Streptococcus pneumoniae vaccine serotypes. The 10 pneumococcal S. pneumoniae vaccine serotypes assessed for this outcome measure were the serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. Pneumococcal ID cases were identified through non-culture pneumococcal diagnostic tests with additional non-culture vaccine type serotyping. Tests used included rapid in-vitro diagnostic tests or Latex agglutination.
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 10211 | 10140
Subjects | 6 | 17

29. Secondary Outcome: Number of Subjects With a First Episode Reported of Invasive Pneumococcal Disease (IPD) Due to Streptococcus (S. pn.) Cross-reactive Pneumococcal Serotypes.
Description: The S. pn. cross-reactive serotypes assessed for this outcome measure were the serotypes 19A, 6A and 9N.
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 10211 | 10140
Subjects | 2 | 1

30. Secondary Outcome: Number of Subjects With a First Episode Reported of Invasive Pneumococcal Disease (IPD) Due to Pneumococcal Serotypes Other Than Streptococcus (S. pn.) Vaccine and Cross-reactive Serotypes.
Description: The serotypes assessed for this outcome measure included among others the pneumococcal serotypes 12F, 16F, 24F, 38 and 8.
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 10211 | 10140
Subjects | 3 | 0

31. Secondary Outcome: Number of Subjects With a First Episode Reported of Invasive Disease (ID) Due to Haemophilus Influenzae
Description: No subject was reported with any case of ID due to Haemophilus influenzae.
Time Frame: Any time from 2 weeks post primary vaccination Dose 3 to study end at Month 22-25
Reporting Status: Not Posted, anticipated posting 2050-12

32. Secondary Outcome: Number of Subjects With Streptococcus Pneumoniae (S. pn.) Vaccine Serotypes Identified in Nasopharyngeal Swabs, in the Carriage Subset.
Description: The 10 pneumococcal S. pn. vaccine serotypes assessed for this outcome measure were the serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. S. pn. serotypes were identified using latex agglutination and by quellung reaction with omni serum. The Carriage Subset consisted in a subgroup of 2,000 subjects enrolled in Panama.
Time Frame: At Months 5, 10-13, 13-16, 14-17, 16-19 and 22-25
Population: The analysis was performed on all vaccinated subjects included in the carriage subset.
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 814 | 814
Subjects
  Month 5 (N=814; 814) | 104 | 123
  Month 10-13 (N=788; 784) | 92 | 123
  Month 13-16 (N=758; 762) | 88 | 109
  Month 14-17 (N=720; 738) | 74 | 103
  Month 16-19 (N=696; 690) | 68 | 98
  Month 22-25 (N=627; 639) | 61 | 86

33. Secondary Outcome: Number of Subjects With Streptococcus Pneumoniae (S. pn.) Cross-reactive Serotypes Identified in Nasopharyngeal Swabs, in the Carriage Subset.
Description: Any serotype belonging to the same serogroup as the Synflorix vaccine serotypes, but different from the vaccine serotypes, was considered for this analysis of carriage S. pn. cross-reactive serotypes. S. pn. serotypes were identified using latex agglutination and by quellung reaction with omni serum. The Carriage Subset consisted in a subgroup of 2,000 subjects enrolled in Panama.
Time Frame: At Months 5, 10-13, 13-16, 14-17, 16-19 and 22-25
Population: The analysis was performed on all vaccinated subjects included in the carriage subset.
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 814 | 814
Subjects
  Month 5 (N=814; 814) | 63 | 67
  Month 10-13 (N=788; 784) | 81 | 63
  Month 13-16 (N=758; 762) | 57 | 63
  Month 14-17 (N=720; 738) | 57 | 49
  Month 16-19 (N=696; 690) | 55 | 57
  Month 22-25 (N=627; 639) | 38 | 46

34. Secondary Outcome: Number of Subjects With Streptococcus Pneumoniae (S. pn.) Serotypes Identified in Nasopharyngeal Swabs Other Than the Synflorix Vaccine and Cross-reactive Serotypes, in the Carriage Subset
Description: S. pn. serotypes were identified using latex agglutination and by quellung reaction with omni serum. The Carriage Subset consisted in a subgroup of 2,000 subjects enrolled in Panama.
Time Frame: At Months 5, 10-13, 13-16, 14-17, 16-19 and 22-25
Population: The analysis was performed on all vaccinated subjects included in the carriage subset.
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 814 | 814
Subjects
  Month 5 (N=814; 814) | 99 | 86
  Month 10-13 (N=788; 784) | 85 | 85
  Month 13-16 (N=758; 762) | 83 | 85
  Month 14-17 (N=720; 738) | 78 | 85
  Month 16-19 (N=696; 690) | 89 | 69
  Month 22-25 (N=627; 639) | 74 | 61

35. Secondary Outcome: Number of Subjects With H. Influenzae Strains Identified in Nasopharyngeal Swabs, in the Carriage Subset
Description: Results included samples confirmed as positive for Haemophilus influenzae (H. influenzae) or non-typeable H. influenzae (NTHi) after differentiation from H. haemolyticus by polymerase chain reaction (PCR) assay. The Carriage Subset contained a subgroup of 2,000 subjects enrolled in Panama.
Time Frame: At Months 5, 10-13, 13-16, 14-17, 16-19 and 22-25
Population: The analysis was performed on all vaccinated subjects included in the carriage subset.
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 824 | 820
Subjects
  Month 5 (N=824; 820) | 36 | 40
  Month 10-13 (N=788;785) | 45 | 44
  Month 13-16 (N=757;762) | 32 | 39
  Month 14-17 (N=720; 737) | 28 | 34
  Month 16-19 (N=696; 690) | 28 | 38
  Month 22-25 (N=628; 640) | 29 | 33

36. Secondary Outcome: Number of Subjects With Acquisition of New Streptococcus Pneumoniae Strains Identified in Nasopharyngeal Swabs, in the Carriage Subset
Description: The Carriage Subset consisted in a subgroup of 2,000 subjects enrolled in Panama.
Time Frame: At Months 10-13, 13-16, 14-17, 16-19 and 22-25
Population: The analysis was performed on all vaccinated subjects included in the carriage subset.
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 788 | 784
Subjects
  Month 10-13 (N=788;784) | 171 | 175
  Month 13-16 (N=758;762) | 145 | 165
  Month 14-17 (N=720;738) | 110 | 137
  Month 16-19 (N=696;690) | 126 | 137
  Month 22-25;N=627;639) | 123 | 124

37. Secondary Outcome: Number of Subjects With Acquisition of New Haemophilus Influenzae Strains Identified in Nasopharyngeal Swabs, in the Carriage Subset.
Description: The Carriage Subset consisted in a subgroup of 2,000 subjects enrolled in Panama.
Time Frame: At Months 10-13, 13-16, 14-17, 16-19 and 22-25
Population: The analysis was performed on all vaccinated subjects included in the carriage subset.
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 788 | 785
Subjects
  Month 10-13 (N=788;785) | 39 | 37
  Month 13-16 (N=757;762) | 27 | 33
  Month 14-17 (N=720;737) | 23 | 28
  Month 16-19 (N=696;690) | 22 | 32
  Month 22-25 (N=628;640) | 28 | 31

38. Secondary Outcome: Number of Subjects With Any Antibiotic Prescription at Least Once During the Entire Study Period, in the Carriage Subset.
Description: The Carriage Subset consisted in a subgroup of 2,000 subjects enrolled in Panama.
Time Frame: Throughout the study (Month 0 to Month 22-25)
Population: The analysis was performed on all vaccinated subjects included in the carriage subset.
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 955 | 966
Subjects | 611 | 626

39. Secondary Outcome: Pneumococcal Antibody Concentrations Against Pneumococcal Vaccine Serotypes, in the Immunogenicity and Tolerability Subset.
Description: Antibody concentrations were measured by 22F enzyme-linked Immunosorbent Assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). Serotypes assessed were the pneumococcal vaccine serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. The cut-off of the assay was >= 0.05 µg/mL. The Immunogenicity and Tolerability Subset included 500 subjects coming from Argentina and Panama respectively.
Time Frame: At Month 5, one month after the third dose of primary vaccination
Population: Analyses were performed on the Primary According-to-Protocol immunogenicity cohort, including all evaluable subjects in the Immunogenicity and Tolerability Subset (500 subjects in Argentina, 500 in Panama) with post primary vaccination assay results against at least 1 study vaccine antigen component and concerning immunogenicity outcomes available.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 334 | 331
µg/mL
  ANTI-1 (N=334;312) | 2.51 [2.29 to 2.75] | 0.04 [0.03 to 0.04]
  ANTI-4 (N=334;328) | 3.26 [2.98 to 3.56] | 0.03 [0.03 to 0.04]
  ANTI-5 (N=334;324) | 4.20 [3.86 to 4.57] | 0.05 [0.04 to 0.05]
  ANITI-6B (N=334;322) | 1.34 [1.18 to 1.52] | 0.03 [0.03 to 0.03]
  ANTI-7F (N=334;330) | 3.86 [3.56 to 4.19] | 0.04 [0.04 to 0.05]
  ANTI-9V (N=334;331) | 3.15 [2.84 to 3.50] | 0.04 [0.03 to 0.04]
  ANTI-14 (N=334;330) | 4.55 [4.07 to 5.10] | 0.09 [0.08 to 0.11]
  ANTI-18C (N=334;328) | 5.32 [4.73 to 5.99] | 0.04 [0.04 to 0.04]
  ANTI-19F (N=334;327) | 5.33 [4.70 to 6.06] | 0.06 [0.05 to 0.07]
  ANTI-23F (N=334;331) | 1.99 [1.76 to 2.26] | 0.04 [0.03 to 0.04]

40. Secondary Outcome: Antibody Concentrations Against Pneumococcal Cross-reactive Serotypes 6A and 19A, in the Immunogenicity and Tolerability Subset
Description: Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). The cut-off of the assay was >= 0.05 µg/mL. The Immunogenicity and Tolerability Subset included 500 subjects coming from Argentina and Panama respectively.
Time Frame: At Month 5, one month after the third dose of primary vaccination
Population: as for outcome 39
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 334 | 326
µg/mL
  ANTI-6A (N=334;321) | 0.32 [0.27 to 0.37] | 0.03 [0.03 to 0.04]
  ANTI-19A (N=334;326) | 0.29 [0.25 to 0.33] | 0.04 [0.04 to 0.05]

41. Secondary Outcome: Antibody Concentrations Against Pneumococcal Vaccine Serotypes, in the Immunogenicity and Tolerability Subset.
Description: as for outcome 39
Time Frame: Before the administration of booster vaccination (PRE), and 1 month and 9 months post booster vaccination (M1 POST-BST and M9 POST-BST)
Population: Analyses were performed on the Booster According-to-Protocol immunogenicity cohort, including all evaluable subjects in the Immunogenicity and Tolerability Subset (500 subjects in Argentina, 500 in Panama) with post booster assay results against at least 1 study vaccine antigen component and concerning immunogenicity outcomes available.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 231 | 214
µg/mL
  ANTI-1, PRE (N=231;203) | 0.35 [0.31 to 0.39] | 0.05 [0.04 to 0.06]
  ANTI-1, M1 POST-BST (N=219;196) | 3.58 [3.15 to 4.07] | 0.06 [0.05 to 0.06]
  ANTI-1, M9 POST-BST (N=206;181) | 0.65 [0.56 to 0.75] | 0.06 [0.05 to 0.06]
  ANTI-4, PRE (N=231;214) | 0.48 [0.42 to 0.55] | 0.04 [0.04 to 0.05]
  ANTI-4, M1 POST-BST (N=217;204) | 6.55 [5.81 to 7.38] | 0.05 [0.04 to 0.05]
  ANTI-4, M9 POST-BST (N=206;183) | 0.87 [0.77 to 0.99] | 0.04 [0.04 to 0.05]
  ANTI-5, PRE (N=231;209) | 0.90 [0.80 to 1.01] | 0.07 [0.07 to 0.09]
  ANTI-5, M1 POST-BST (N=219;199) | 5.73 [5.04 to 6.50] | 0.07 [0.06 to 0.08]
  ANTI-5, M9 POST-BST (N=206;182) | 1.19 [1.05 to 1.36] | 0.09 [0.08 to 0.10]
  ANTI-6B, PRE (N=229;212) | 0.55 [0.47 to 0.64] | 0.04 [0.03 to 0.04]
  ANTI-6B, M1 POST-BST (N=217;198) | 3.32 [2.92 to 3.77] | 0.04 [0.03 to 0.04]
  ANTI-6B, M9 POST-BST (N=206;182) | 0.83 [0.71 to 0.96] | 0.05 [0.04 to 0.06]
  ANTI-7F, PRE (N=231;210) | 0.94 [0.84 to 1.04] | 0.06 [0.05 to 0.07]
  ANTI-7F, M1 POST-BST (N=218;198) | 5.77 [5.23 to 6.36] | 0.06 [0.05 to 0.07]
  ANTI-7F, M9 POST-BST (N=206;182) | 1.32 [1.19 to 1.45] | 0.07 [0.05 to 0.08]
  ANTI-9V, PRE (N=230;214) | 1.14 [1.00 to 1.31] | 0.04 [0.04 to 0.05]
  ANTI-9V, M1 POST-BST (N=218;203) | 7.34 [6.51 to 8.27] | 0.04 [0.04 to 0.05]
  ANTI-9V, M9 POST-BST (N=206;182) | 1.80 [1.59 to 2.03] | 0.05 [0.04 to 0.06]
  ANTI-14, PRE (N=231;214) | 1.15 [1.15 to 1.35] | 0.11 [0.09 to 0.13]
  ANTI-14, M1 POST-BST (N=219;200) | 9.31 [8.18 to 10.60] | 0.12 [0.10 to 0.14]
  ANTI-14, M9 POST-BST (N=206;183) | 1.98 [1.74 to 2.26] | 0.17 [0.14 to 0.21]
  ANTI-18C, PRE (N=231;210) | 0.90 [0.79 to 1.03] | 0.05 [0.04 to 0.06]
  ANTI-18C, M1 POST-BST (N=219;203) | 16.38 [14.47 to 18.55] | 0.05 [0.04 to 0.05]
  ANTI-18C, M9 POST-BST (N=206;181) | 2.50 [2.21 to 2.83] | 0.05 [0.04 to 0.06]
  ANTI-19F, PRE (N=231;206) | 1.27 [1.09 to 1.48] | 0.06 [0.05 to 0.07]
  ANTI-19F, M1 POST-BST (N=219;198) | 9.40 [8.40 to 10.52] | 0.07 [0.05 to 0.08]
  ANTI-19F, M9 POST-BST (N=205;181) | 2.47 [2.16 to 2.84] | 0.10 [0.08 to 0.12]
  ANTI-23F, PRE (N=229;204) | 0.62 [0.53 to 0.72] | 0.04 [0.03 to 0.05]
  ANTI-23F, M1 POST-BST (N=218;201) | 4.02 [3.49 to 4.62] | 0.04 [0.03 to 0.04]
  ANTI-23F, M9 POST-BST (N=206;179) | 0.92 [0.80 to 1.06] | 0.05 [0.04 to 0.06]

42. Secondary Outcome: Antibody Concentrations Against Pneumococcal Cross-reactive Serotypes 6A and 19A, in the Immunogenicity and Tolerability Subset
Description: as for outcome 40
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 231 | 214
µg/mL
  ANTI-6A, PRE (N=231;214) | 0.22 [0.18 to 0.26] | 0.04 [0.04 to 0.05]
  ANTI-6A, M1 POST-BST (N=219;204) | 1.14 [0.93 to 1.40] | 0.04 [0.03 to 0.04]
  ANTI-6A, M9 POST-BST (N=206;183) | 0.31 [0.26 to 0.37] | 0.05 [0.04 to 0.06]
  ANTI-19A, PRE (N=229;212) | 0.25 [0.21 to 0.30] | 0.05 [0.05 to 0.07]
  ANTI-19A, M1 POST-BST (N=218;201) | 1.34 [1.11 to 1.62] | 0.06 [0.05 to 0.07]
  ANTI-19A, M9 POST-BST (N=206;181) | 0.54 [0.46 to 0.65] | 0.09 [0.07 to 0.11]

43. Secondary Outcome: Number of Subjects With Antibody Concentrations Against Pneumococcal Vaccine Serotypes >= 0.20 Micrograms Per Milliliter (µg/mL), in the Immunogenicity and Tolerability Subset
Description: Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA). Serotypes assessed were the pneumococcal vaccine serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. The Immunogenicity and Tolerability Subset included 500 subjects coming from Argentina and Panama respectively.
Time Frame: At Month 5, one month after the third dose of primary vaccination
Population: as for outcome 39
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 334 | 331
Subjects
  ANTI-1 (N=334;312) | 333 | 13
  ANTI-4 (N=334;328) | 332 | 11
  ANTI-5 (N=334;324) | 333 | 22
  ANITI-6B (N=334;322) | 311 | 8
  ANTI-7F (N=334;330) | 333 | 28
  ANTI-9V (N=334;331) | 330 | 19
  ANTI-14 (N=334;330) | 328 | 77
  ANTI-18C (N=334;328) | 330 | 21
  ANTI-19F (N=334;327) | 325 | 40
  ANTI-23F (N=334;331) | 321 | 15

44. Secondary Outcome: Number of Subjects With Antibody Concentrations Against Pneumococcal Cross-reactive Serotypes 6A and 19A >= 0.20 Micrograms Per Milliliter (µg/mL), in the Immunogenicity and Tolerability Subset
Description: Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA). The Immunogenicity and Tolerability Subset included 500 subjects coming from Argentina and Panama respectively.
Time Frame: At Month 5, one month after the third dose of primary vaccination
Population: as for outcome 39
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 334 | 326
Subjects
  ANTI-6A (N=334;321) | 215 | 5
  ANTI-19A (N=334;326) | 204 | 18

45. Secondary Outcome: Number of Subjects With Antibody Concentrations Against Pneumococcal Vaccine Serotypes >= 0.20 Micrograms Per Milliliter (µg/mL), in the Immunogenicity and Tolerability Subset
Description: Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA). Serotypes assessed with the pneumococcal vaccine serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. The Immunogenicity and Tolerability Subset included 500 subjects coming from Argentina and Panama respectively.
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 231 | 214
Subjects
  ANTI-1, PRE (N=231;203) | 164 | 14
  ANTI-1, M1 POST-BST (N=219;196) | 219 | 19
  ANTI-1, M9 POST-BST (N=206;181) | 186 | 14
  ANTI-4, PRE (N=231;214) | 190 | 26
  ANTI-4, M1 POST-BST (N=217;204) | 217 | 24
  ANTI-4, M9 POST-BST (N=206;183) | 198 | 15
  ANTI-5, PRE (N=231;209) | 218 | 27
  ANTI-5, M1 POST-BST (N=219;199) | 219 | 30
  ANTI-5, M9 POST-BST (N=206;182) | 200 | 34
  ANTI-6B, PRE (N=229;212) | 182 | 12
  ANTI-6B, M1 POST-BST (N=217;198) | 215 | 13
  ANTI-6B, M9 POST-BST (N=206;182) | 192 | 21
  ANTI-7F, PRE (N=231;210) | 222 | 34
  ANTI-7F, M1 POST-BST (N=218;198) | 218 | 36
  ANTI-7F, M9 POST-BST (N=206;182) | 205 | 31
  ANTI-9V, PRE (N=230;214) | 221 | 22
  ANTI-9V, M1 POST-BST (N=218;203) | 218 | 14
  ANTI-9V, M9 POST-BST (N=206;182) | 206 | 26
  ANTI-14, PRE (N=231;214) | 217 | 51
  ANTI-14, M1 POST-BST (N=219;200) | 219 | 52
  ANTI-14, M9 POST-BST (N=206;183) | 204 | 68
  ANTI-18C, PRE (N=231;210) | 217 | 22
  ANTI-18C, M1 POST-BST (N=219;203) | 219 | 21
  ANTI-18C, M9 POST-BST (N=206;181) | 205 | 18
  ANTI-19F, PRE (N=231;206) | 221 | 35
  ANTI-19F, M1 POST-BST (N=219;198) | 218 | 39
  ANTI-19F, M9 POST-BST (N=205;181) | 204 | 52
  ANTI-23F, PRE (N=229;204) | 198 | 15
  ANTI-23F, M1 POST-BST (N=218;201) | 216 | 14
  ANTI-23F, M9 POST-BST (N=206;179) | 196 | 25

46. Secondary Outcome: Number of Subjects With Pneumococcal Antibody Concentrations Against Cross-reactive Serotypes 6A and 19A Higher >= 0.20 Micrograms Per Milliliter (µg/mL), in the Immunogenicity and Tolerability Subset
Description: as for outcome 44
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 231 | 214
Subjects
  ANTI-6A, PRE (N=231;214) | 119 | 14
  ANTI-6A, M1 POST-BST (N=219;204) | 187 | 12
  ANTI-6A, M9 POST-BST (N=206;183) | 129 | 24
  ANTI-19A, PRE (N=229;212) | 131 | 28
  ANTI-19A, M1 POST-BST (N=218;201) | 197 | 27
  ANTI-19A, M9 POST-BST (N=206;181) | 165 | 47

47. Secondary Outcome: Number of Subjects With Antibody Concentrations Against Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F >= 0.05 Microgram Per Milliliter (µg/mL), in the Immunogenicity and Tolerability Subset
Description: A seropositive subject was defined as a subject with antibody concentrations against vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F => 0.05 µg/mL. The Immunogenicity and Tolerability Subset included 500 subjects coming from Argentina and Panama respectively.
Time Frame: At Month 5, one month after the third dose of primary vaccination
Population: as for outcome 39
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 334 | 331
Subjects
  ANTI-1 (N=334;312) | 333 | 88
  ANTI-4 (N=334;328) | 333 | 48
  ANTI-5 (N=334;324) | 334 | 153
  ANITI-6B (N=334;322) | 324 | 48
  ANTI-7F (N=334;330) | 333 | 116
  ANTI-9V (N=334;331) | 331 | 68
  ANTI-14 (N=334;330) | 333 | 234
  ANTI-18C (N=334;328) | 333 | 92
  ANTI-19F (N=334;327) | 331 | 176
  ANTI-23F (N=334;331) | 328 | 78

48. Secondary Outcome: Number of Subjects With Pneumococcal Antibody Concentrations Against Serotypes 6A and 19A >= 0.05 µg/mL, in the Immunogenicity and Tolerability Subset
Description: A seropositive subject was defined as a subject with antibody concentrations against cross-reactive pneumococcal serotypes 6A and 19A>= 0.05 µg/mL. The Immunogenicity and Tolerability Subset included 500 subjects coming from Argentina and Panama respectively.
Time Frame: At Month 5, one month after the third dose of primary vaccination
Population: as for outcome 39
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 334 | 326
Subjects
  ANTI-6A (N=334;321) | 306 | 77
  ANTI-19A (N=334;326) | 303 | 120

49. Secondary Outcome: Number of Subjects With Antibody Concentrations Against Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F >= 0.05 Microgram Per Milliliter (µg/mL), in the Immunogenicity and Tolerability Subset
Description: as for outcome 47
Time Frame: Before the administration of booster vaccination (PRE), and 1 month and 9 months post booster vaccination (M1 POST-BST and M9 POST-BST
Population: as for outcome 41
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 231 | 214
Subjects
  ANTI-1, PRE (N=231;203) | 231 | 87
  ANTI-1, M1 POST-BST (N=219;196) | 219 | 101
  ANTI-1, M9 POST-BST (N=206;181) | 206 | 95
  ANTI-4, PRE (N=231;214) | 231 | 52
  ANTI-4, M1 POST-BST (N=217;204) | 217 | 65
  ANTI-4, M9 POST-BST (N=206;183) | 206 | 58
  ANTI-5, PRE (N=231;209) | 231 | 150
  ANTI-5, M1 POST-BST (N=219;199) | 219 | 142
  ANTI-5, M9 POST-BST (N=206;182) | 206 | 133
  ANTI-6B, PRE (N=229;212) | 226 | 60
  ANTI-6B, M1 POST-BST (N=217;198) | 216 | 54
  ANTI-6B, M9 POST-BST (N=206;182) | 206 | 72
  ANTI-7F, PRE (N=231;210) | 231 | 79
  ANTI-7F, M1 POST-BST (N=218;198) | 218 | 79
  ANTI-7F, M9 POST-BST (N=206;182) | 206 | 87
  ANTI-9V, PRE (N=230;214) | 230 | 51
  ANTI-9V, M1 POST-BST (N=218;203) | 218 | 58
  ANTI-9V, M9 POST-BST (N=206;182) | 206 | 68
  ANTI-14, PRE (N=231;214) | 231 | 157
  ANTI-14, M1 POST-BST (N=219;200) | 219 | 160
  ANTI-14, M9 POST-BST (N=206;183) | 206 | 154
  ANTI-18C, PRE (N=231;210) | 230 | 72
  ANTI-18C, M1 POST-BST (N=219;203) | 219 | 71
  ANTI-18C, M9 POST-BST (N=206;181) | 206 | 73
  ANTI-19F, PRE (N=231;206) | 231 | 71
  ANTI-19F, M1 POST-BST (N=219;198) | 219 | 85
  ANTI-19F, M9 POST-BST (N=205;181) | 205 | 93
  ANTI-23F, PRE (N=229;204) | 223 | 44
  ANTI-23F, M1 POST-BST (N=218;201) | 216 | 44
  ANTI-23F, M9 POST-BST (N=206;179) | 206 | 62

50. Secondary Outcome: Number of Subjects With Pneumococcal Antibody Concentrations Against Serotypes 6A and 19A >= 0.05 µg/mL, in the Immunogenicity and Tolerability Subset
Description: as for outcome 48
Time Frame: Before the administration of booster vaccination (PRE), and 1 month and 9 months post booster vaccination (M1 POST-BST and M9 POST-BST) .
Population: as for outcome 41
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 231 | 214
Subjects
  ANTI-6A, PRE (N=231;214) | 210 | 61
  ANTI-6A, M1 POST-BST (N=219;204) | 214 | 61
  ANTI-6A, M9 POST-BST (N=206;183) | 196 | 69
  ANTI-19A, PRE (N=229;212) | 208 | 76
  ANTI-19A, M1 POST-BST (N=218;201) | 212 | 83
  ANTI-19A, M9 POST-BST (N=206;181) | 201 | 89

51. Secondary Outcome: Titers for Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F, in the Immunogenicity and Tolerability Subset
Description: The cut-off of the assay was >= 8. The Immunogenicity and Tolerability Subset included 500 subjects coming from Argentina and Panama respectively.
Time Frame: At Month 5, one month after the third dose of primary vaccination,
Population: as for outcome 39
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 317 | 317
Titers
  OPSONO-1 (N=306;305) | 139.5 [116.8 to 166.5] | 4.8 [4.5 to 5.3]
  OPSONO-4 (N=310;299) | 771.7 [686.5 to 867.6] | 5.1 [4.5 to 5.8]
  OPSONO-5 (N=313;314) | 224.8 [196.0 to 257.8] | 4.5 [4.2 to 4.8]
  OPSONO-6B (N=315;309) | 689.7 [553.2 to 859.7] | 5.4 [4.6 to 6.2]
  OPSONO-7F (N=302;266) | 4656.7 [4175.6 to 5193.3] | 110.4 [78.8 to 154.7]
  OPSONO-9V (N=312;302) | 1690.4 [1489.4 to 1918.7] | 14.6 [11.6 to 18.2]
  OPSONO-14 (N=308;273) | 908.5 [795.2 to 1038.1] | 16.5 [12.9 to 21.1]
  OPSONO-18C (N=308;317) | 310.9 [259.4 to 372.6] | 4.4 [4.1 to 4.7]
  OPSONO-19F (N=304;314) | 383.0 [308.5 to 475.5] | 4.7 [4.3 to 5.2]
  OPSONO-23F (N=317;282) | 2167.4 [1863.4 to 2521.1] | 14.5 [11.0 to 19.1]

52. Secondary Outcome: Titers for Opsonophagocytic Activity Against Cross-reactive Pneumococcal Serotypes 6A and 19A, in the Immunogenicity and Tolerability Subset
Description: as for outcome 51
Time Frame: At Month 5, one month after the third dose of primary vaccination
Population: Analyses were performed on the Primary According-to-Protocol immunogenicity cohort, including all evaluable subjects in the Immunogenicity and Safety Subset (500 subjects in Argentina, 500 in Panama) with post primary vaccination assay results against at least 1 study vaccine antigen component and concerning immunogenicity outcomes available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 302 | 309
Titers
  OPSONO-6A (N=297;305) | 156.9 [121.8 to 202.1] | 5.0 [4.5 to 5.5]
  OPSONO-19A (N=302;309) | 18.2 [14.5 to 22.9] | 4.1 [4.0 to 4.3]

53. Secondary Outcome: Titers for Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F, in the Immunogenicity and Tolerability Subset
Description: as for outcome 51
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 221 | 210
Titers
  OPSONO-1, PRE (N=221;210) | 9.0 [7.4 to 10.9] | 4.6 [4.2 to 5.0]
  OPSONO-1, M1 POST-BST (N=209;200) | 357.5 [281.8 to 453.5] | 4.8 [4.4 to 5.4]
  OPSONO-1, M9 POST-BST (N=196;176) | 34.4 [26.6 to 44.7] | 4.6 [4.2 to 5.1]
  OPSONO-4, PRE (N=208;193) | 29.2 [21.2 to 40.2] | 8.6 [6.4 to 11.5]
  OPSONO-4, M1 POST-BST (N=207;193) | 2853.5 [2365.5 to 3442.1] | 8.3 [6.3 to 10.9]
  OPSONO-4, M9 POST-BST (N=192;173) | 165.6 [115.3 to 237.9] | 8.1 [6.1 to 10.8]
  OPSONO-5, PRE (N=205;204) | 18.5 [15.4 to 22.3] | 4.3 [4.1 to 4.6]
  OPSONO-5, M1 POST-BST (N=196;187) | 306.1 [252.0 to 371.8] | 4.4 [4.1 to 4.7]
  OPSONO-5, M9 POST-BST (N=192;173) | 44.1 [35.5 to 54.7] | 4.2 [4.0 to 4.4]
  OPSONO-6B, PRE (N=209;197) | 95.5 [70.1 to 130.1] | 7.6 [6.0 to 9.8]
  OPSONO-6B, M1 POST-BST (N=203;190) | 1123.4 [939.2 to 1343.9] | 7.1 [5.6 to 8.9]
  OPSONO-6B, M9 POST-BST (N=178;165) | 128.9 [92.7 to 179.2] | 11.4 [8.3 to 15.8]
  OPSONO-7F, PRE (N=217;202) | 1522.8 [1338.5 to 1732.6] | 979.5 [821.2 to 1168.5]
  OPSONO-7F, M1 POST-BST (N=205;196) | 4336.3 [3607.9 to 5211.8] | 746.4 [590.7 to 943.1]
  OPSONO-7F, M9 POST-BST (N=192;172) | 2598.0 [2232.0 to 3024.1] | 1214.3 [1011.4 to 1458.0]
  OPSONO-9V, PRE (N=213;188) | 709.4 [601.7 to 836.3] | 233.7 [175.3 to 311.4]
  OPSONO-9V, M1 POST-BST (N=200;189) | 3763.0 [3317.5 to 4268.3] | 250.9 [186.1 to 338.4]
  OPSONO-9V, M9 POST-BST (N=194;168) | 1320.3 [1153.1 to 1511.7] | 337.4 [252.4 to 451.0]
  OPSONO-14, PRE (N=205;192) | 121.2 [89.7 to 163.8] | 27.0 [18.9 to 38.5]
  OPSONO-14, M1 POST-BST (N=209;188) | 2659.6 [2266.2 to 3121.3] | 21.7 [15.0 to 31.2]
  OPSONO-14, M9 POST-BST (N=185;159) | 330.6 [242.7 to 450.5] | 27.6 [18.3 to 41.8]
  OPSONO-18C, PRE (N=204;191) | 15.0 [11.5 to 19.6] | 4.8 [4.2 to 5.4]
  OPSONO-18C, M1 POST-BST (N=188;187) | 2426.0 [2041.8 to 2882.5] | 5.2 [4.4 to 6.0]
  OPSONO-18C, M9 POST-BST (N=170;164) | 722.0 [553.6 to 941.6] | 5.3 [4.4 to 6.5]
  OPSONO-19F, PRE (N=218;205) | 24.3 [19.6 to 30.1] | 5.0 [4.4 to 5.7]
  OPSONO-19F, M1 POST-BST (N=199;200) | 657.5 [497.4 to 869.1] | 5.0 [4.4 to 5.7]
  OPSONO-19F, M9 POST-BST (N=194;170) | 118.0 [90.6 to 153.7] | 4.8 [4.3 to 5.4]
  OPSONO-23F, PRE (N=215;199) | 679.3 [494.3 to 933.6] | 76.9 [49.0 to 120.6]
  OPSONO-23F, M1 POST-BST (N=206;190) | 4278.3 [3609.3 to 5071.3] | 99.7 [62.7 to 158.6]
  OPSONO-23F, M9 POST-BST (N=187;167) | 999.6 [711.8 to 1403.9] | 109.4 [65.7 to 182.2]

54. Secondary Outcome: Titers for Opsonophagocytic Activity Against Pneumococcal Serotypes 6A and 19A in the Immunogenicity and Tolerability Subset
Description: as for outcome 51
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 217 | 204
Titers
  OPSONO-6A, PRE (N=189;194) | 43.8 [31.0 to 62.0] | 7.1 [5.7 to 8.9]
  OPSONO-6A, M1 POST BST (N=185;185) | 277.2 [198.7 to 386.7] | 7.6 [6.0 to 9.7]
  OPSONO-6A, M9 POST-BST (N=175;156) | 63.9 [44.3 to 92.0] | 17.2 [12.1 to 24.4]
  OPSONO-19A, PRE (N=217;204) | 6.3 [5.3 to 7.4] | 5.0 [4.4 to 5.6]
  OPSONO-19A, M1 POST-BST (N=200;197) | 132.8 [97.5 to 180.8] | 5.4 [4.7 to 6.2]
  OPSONO-19A, M9 POST-BST (N=187;171) | 26.1 [19.5 to 35.1] | 6.3 [5.3 to 7.5]

55. Secondary Outcome: Number of Subjects With Titers for Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F => 8, in the Immunogenicity and Tolerability Subset
Description: A seropositive subject was defined as a subject with titers for opsonophagocytic activity against vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F >= 8. The Immunogenicity and Tolerability Subset included 500 subjects coming from Argentina and Panama respectively.
Time Frame: At Month 5, one month after the third dose of primary vaccination
Population: as for outcome 39
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 317 | 317
Subjects
  OPSONO-1 (N=306;305) | 280 | 25
  OPSONO-4 (N=310;299) | 306 | 15
  OPSONO-5 (N=313;314) | 303 | 13
  OPSONO-6B (N=315;309) | 286 | 16
  OPSONO-7F (N=302;266) | 302 | 162
  OPSONO-9V (N=312;302) | 311 | 98
  OPSONO-14 (N=308;273) | 306 | 95
  OPSONO-18C (N=308;317) | 290 | 8
  OPSONO-19F (N=304;314) | 277 | 16
  OPSONO-23F (N=317;282) | 311 | 68

56. Secondary Outcome: Number of Subjects With Titers for Opsonophagocytic Activity Against Cross-reactive Pneumococcal Serotypes 6A and 19A >= 8, in the Immunogenicity and Tolerability Subset
Description: A seropositive subject was defined as a subject with titers for opsonophagocytic activity against cross-reactive pneumococcal serotypes 6A and 19A >= 8. The Immunogenicity and Tolerability Subset included 500 subjects coming from Argentina and Panama respectively.
Time Frame: At Month 5, one month after the third dose of primary vaccination
Population: as for outcome 39
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 302 | 309
Subjects
  OPSONO-6A (N=297;305) | 232 | 16
  OPSONO-19A (N=302;309) | 121 | 5

57. Secondary Outcome: Number of Subjects With Titers for Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F >= 8, in the Immunogenicity and Tolerability Subset
Description: as for outcome 55
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 221 | 210
Subjects
  OPSONO-1, PRE (N=221;210) | 58 | 9
  OPSONO-1, M1 POST-BST (N=209;200) | 195 | 14
  OPSONO-1, M9 POST-BST (N=196;176) | 127 | 10
  OPSONO-4, PRE (N=208;193) | 108 | 25
  OPSONO-4, M1 POST-BST (N=207;193) | 206 | 26
  OPSONO-4, M9 POST-BST (N=192;173) | 147 | 22
  OPSONO-5, PRE (N=205;204) | 138 | 7
  OPSONO-5, M1 POST-BST (N=196;187) | 194 | 10
  OPSONO-5, M9 POST-BST (N=192;173) | 157 | 3
  OPSONO-6B, PRE (N=209;197) | 162 | 27
  OPSONO-6B, M1 POST-BST (N=203;190) | 200 | 23
  OPSONO-6B, M9 POST-BST (N=178;165) | 146 | 35
  OPSONO-7F, PRE (N=217;202) | 217 | 197
  OPSONO-7F, M1 POST-BST (N=205;196) | 203 | 185
  OPSONO-7F, M9 POST-BST (N=192;172) | 192 | 169
  OPSONO-9V, PRE (N=213;188) | 212 | 159
  OPSONO-9V, M1 POST-BST (N=200;189) | 200 | 157
  OPSONO-9V, M9 POST-BST (N=194;168) | 194 | 148
  OPSONO-14, PRE (N=205;192) | 158 | 73
  OPSONO-14, M1 POST-BST (N=209;188) | 208 | 61
  OPSONO-14, M9 POST-BST (N=185;159) | 160 | 57
  OPSONO-18C, PRE (N=204;191) | 86 | 8
  OPSONO-18C, M1 POST-BST (N=188;187) | 187 | 11
  OPSONO-18C, M9 POST-BST (N=170;164) | 165 | 10
  OPSONO-19F, PRE (N=218;205) | 150 | 14
  OPSONO-19F, M1 POST-BST (N=199;200) | 186 | 13
  OPSONO-19F, M9 POST-BST (N=194;170) | 168 | 11
  OPSONO-23F, PRE (N=215;199) | 190 | 94
  OPSONO-23F, M1 POST-BST (N=206;190) | 205 | 97
  OPSONO-23F, M9 POST-BST (N=187;167) | 167 | 85

58. Secondary Outcome: Number of Subjects With Titers for Opsonophagocytic Activity Against Pneumococcal Cross-reactive Serotypes 6A and 19A >= 8, in the Immunogenicity and Tolerability Subset
Description: A seropositive subject was a subject with titers for opsonophagocytic activity against pneumococcal cross-reactive serotypes 6A and 19A >= 8. The Immunogenicity and Tolerability Subset included 500 subjects coming from Argentina and Panama respectively.
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 217 | 204
Subjects
  OPSONO-6A, PRE (N=189;194) | 99 | 24
  OPSONO-6A, M1 POST BST (N=185;185) | 150 | 26
  OPSONO-6A, M9 POST-BST (N=175;156) | 104 | 50
  OPSONO-19A, PRE (N=217;204) | 32 | 14
  OPSONO-19A, M1 POST-BST (N=200;197) | 161 | 20
  OPSONO-19A, M9 POST-BST (N=187;171) | 108 | 32

59. Secondary Outcome: Concentrations of Antibodies Against Protein D (ANTI-PD), in the Immunogenicity and Tolerability Subset
Description: ANTI-PD concentrations are expressed as geometric mean concentrations (GMCs), in enzyme-linked immunosorbent assay (ELISA) unit per milliliter (EL.U/mL). The Immunogenicity and Tolerability Subset included 500 subjects coming from Argentina and Panama respectively.
Time Frame: At Month 5, one month after the third dose of primary vaccination
Population: as for outcome 39
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 334 | 325
EL.U/mL | 2455.2 [2248.3 to 2681.1] | 101.2 [91.3 to 112.2]

60. Secondary Outcome: Concentrations of Antibodies Against Protein D (ANTI-PD), in the Immunogenicity and Tolerability Subset
Description: as for outcome 59
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 230 | 211
EL.U/mL
  ANTI-PD, PRE (N=230;211) | 638.6 [556.2 to 733.2] | 103.1 [90.5 to 117.5]
  ANTI-PD, M1 POST BST (N=218;195) | 2787.0 [2435.9 to 3188.7] | 92.4 [82.6 to 103.3]
  ANTI-PD, M9 POST-BST (N=206;182) | 824.1 [704.2 to 964.4] | 94.5 [84.4 to 105.8]

61. Secondary Outcome: Number of Subjects With Anti-protein D (ANTI-PD) Antibody Concentrations >= 100 Enzyme-linked Immunosorbent Assay Units Per Milliliter ( EL.U/mL), in the Immunogenicity and Tolerability Subset
Description: A seropositive subject was defined as a subject with ANTI-PD antibody concentrations >= 100 EL.U/mL. The Immunogenicity and Tolerability Subset included 500 subjects coming from Argentina and Panama respectively.
Time Frame: At Month 5, one month after the third dose of primary vaccination
Population: as for outcome 39
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 334 | 325
Subjects | 333 | 141

62. Secondary Outcome: Number of Subjects With Anti-protein D (ANTI-PD) Antibody Concentrations >= 100 Enzyme-linked Immunosorbent Assay Units Per Milliliter ( EL.U/mL), in the Immunogenicity and Tolerability Subset.
Description: as for outcome 61
Time Frame: as for outcome 49
Population: Analyses were performed on the Booster According-to-Protocol immunogenicity cohort, including all evaluable subjects in the Immunogenicity and Safety Subset (500 subjects in Argentina, 500 in Panama) with post booster assay results against at least 1 study vaccine antigen component and concerning immunogenicity outcomes available.
Measure: Number; unit: Subjects
Arm/Group | Synflorix Group | Control Group
Number analyzed (Participants) | 230 | 211
Subjects
  ANTI-PD, PRE (N=230;211) | 223 | 96
  ANTI-PD, M1 POST BST (N=218;195) | 218 | 83
  ANTI-PD, M9 POST-BST (N=206;182) | 198 | 84

ADVERSE EVENTS:
Time Frame: SAEs and unsolicited AEs: throughout the study (Months 0 to 22-25). Solicited symptoms: 4-day follow-up period across the 3 doses of primary study vaccine course/ 4-day follow-up period post booster vaccination. Reports for SAEs were collected from all subjects from the Total Vaccinated cohort (TVC). Reports for unsolicited AEs and for solicited symptoms were collected from subjects from the Panama Subset and from the Immunogenicity and Tolerability Subset, respectively.
Description: For this study, the Total Number (#) of Participants Affected by Other (non-serious) Adverse Events (AEs) was analyzed separately for expected AEs and for unexpected AEs. A consolidated analysis of all expected and unexpected AEs was not technically possible to be performed and the relevant data are no longer available. Therefore, the Total #Participants Affected in Other Adverse Events Table is currently populated by the highest value of #Participants affected within other AE's table.
Arm/Group | Synflorix Group | Control Group
All-Cause Mortality (participants affected / at risk) | 19/11798 | 26/11799
Serious Adverse Events (participants affected / at risk) | 2534/11798 | 2668/11799
Other Adverse Events (participants affected / at risk) | 3530/3602 | 3518/3612
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix Group (N=11798) | Control Group (N=11799)
Anaemia (Blood and lymphatic system disorders) | 5 | 9
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 4
Haemolysis (Blood and lymphatic system disorders) | 1 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 1
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 2 | 1
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 | 0
Hypersplenism (Blood and lymphatic system disorders) | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 3 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukaemoid reaction (Blood and lymphatic system disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 12 | 19
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Cyanosis (Cardiac disorders) | 1 | 1
Intracardiac mass (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Cerebral palsy (Congenital, familial and genetic disorders) | 0 | 1
Coarctation of the aorta (Congenital, familial and genetic disorders) | 0 | 1
Congenital absence of bile ducts (Congenital, familial and genetic disorders) | 1 | 0
Congenital oral malformation (Congenital, familial and genetic disorders) | 0 | 1
Congenital syphilis (Congenital, familial and genetic disorders) | 1 | 0
Cystic fibrosis (Congenital, familial and genetic disorders) | 3 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 1 | 0
Heart disease congenital (Congenital, familial and genetic disorders) | 0 | 1
Laryngomalacia (Congenital, familial and genetic disorders) | 1 | 0
Meningomyelocele (Congenital, familial and genetic disorders) | 1 | 0
Porencephaly (Congenital, familial and genetic disorders) | 0 | 1
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 | 1
Retinoblastoma (Congenital, familial and genetic disorders) | 1 | 0
Sickle cell anaemia (Congenital, familial and genetic disorders) | 1 | 1
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 0 | 2
Spinal muscular atrophy (Congenital, familial and genetic disorders) | 1 | 0
Thalassaemia sickle cell (Congenital, familial and genetic disorders) | 0 | 1
Hyperadrenalism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal mass (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 5
Acute abdomen (Gastrointestinal disorders) | 2 | 0
Appendix disorder (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 11 | 10
Diarrhoea (Gastrointestinal disorders) | 63 | 53
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 15 | 20
Faecaloma (Gastrointestinal disorders) | 2 | 3
Food poisoning (Gastrointestinal disorders) | 5 | 1
Gastritis (Gastrointestinal disorders) | 1 | 4
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 3
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 4 | 3
Ileus paralytic (Gastrointestinal disorders) | 33 | 23
Infantile colic (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 3
Inguinal hernia, obstructive (Gastrointestinal disorders) | 5 | 3
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 14 | 11
Malabsorption (Gastrointestinal disorders) | 0 | 1
Mallory-weiss syndrome (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 6
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 42 | 37
Crying (General disorders) | 1 | 1
Effusion (General disorders) | 1 | 0
Electrocution (General disorders) | 2 | 2
Hypothermia (General disorders) | 1 | 1
Multi-organ failure (General disorders) | 1 | 0
Pyrexia (General disorders) | 24 | 31
Sudden death (General disorders) | 0 | 1
Sudden infant death syndrome (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 2 | 0
Food allergy (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 5 | 6
Immunodeficiency (Immune system disorders) | 0 | 1
Milk allergy (Immune system disorders) | 0 | 1
Selective iga immunodeficiency (Immune system disorders) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 11 | 9
Abscess limb (Infections and infestations) | 10 | 16
Abscess neck (Infections and infestations) | 4 | 8
Abscess of eyelid (Infections and infestations) | 1 | 0
Acarodermatitis (Infections and infestations) | 0 | 1
Acquired immunodeficiency syndrome (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 2 | 3
Adenoiditis (Infections and infestations) | 1 | 4
Adenovirus infection (Infections and infestations) | 0 | 1
Amoebiasis (Infections and infestations) | 0 | 2
Amoebic dysentery (Infections and infestations) | 0 | 3
Anal abscess (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 3 | 3
Appendicitis perforated (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 3 | 2
Ascariasis (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 14 | 12
Bacteraemia (Infections and infestations) | 4 | 6
Bacterial diarrhoea (Infections and infestations) | 2 | 2
Bacterial infection (Infections and infestations) | 0 | 2
Breast abscess (Infections and infestations) | 0 | 1
Bronchiolitis (Infections and infestations) | 473 | 518
Bronchitis (Infections and infestations) | 124 | 129
Bronchopneumonia (Infections and infestations) | 106 | 95
Bullous impetigo (Infections and infestations) | 1 | 0
Burn infection (Infections and infestations) | 2 | 1
Cat scratch disease (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 45 | 46
Cellulitis of male external genital organ (Infections and infestations) | 1 | 1
Cellulitis orbital (Infections and infestations) | 1 | 1
Colostomy infection (Infections and infestations) | 1 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 1
Conjunctivitis chlamydial (Infections and infestations) | 0 | 1
Conjunctivitis infective (Infections and infestations) | 1 | 0
Croup infectious (Infections and infestations) | 10 | 7
Cytomegalovirus hepatitis (Infections and infestations) | 1 | 1
Dengue fever (Infections and infestations) | 18 | 15
Diarrhoea infectious (Infections and infestations) | 2 | 0
Dysentery (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 1 | 2
Empyema (Infections and infestations) | 2 | 2
Encephalitis viral (Infections and infestations) | 1 | 1
Enteritis infectious (Infections and infestations) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 4 | 2
Exanthema subitum (Infections and infestations) | 4 | 4
External ear cellulitis (Infections and infestations) | 2 | 0
Fungal skin infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 553 | 497
Gastroenteritis adenovirus (Infections and infestations) | 1 | 3
Gastroenteritis bacterial (Infections and infestations) | 8 | 9
Gastroenteritis rotavirus (Infections and infestations) | 38 | 49
Gastroenteritis shigella (Infections and infestations) | 8 | 8
Gastroenteritis viral (Infections and infestations) | 9 | 9
Giardiasis (Infections and infestations) | 1 | 3
Gingivitis (Infections and infestations) | 0 | 1
Hantaviral infection (Infections and infestations) | 1 | 0
Herpangina (Infections and infestations) | 2 | 0
Herpes simplex (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1
Impetigo (Infections and infestations) | 10 | 4
Infected bites (Infections and infestations) | 0 | 1
Infected cyst (Infections and infestations) | 2 | 0
Infected fistula (Infections and infestations) | 0 | 1
Infectious mononucleosis (Infections and infestations) | 5 | 4
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 2
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 9 | 14
Lobar pneumonia (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Lymph node abscess (Infections and infestations) | 2 | 0
Mastoiditis (Infections and infestations) | 2 | 0
Meningitis (Infections and infestations) | 1 | 2
Meningitis aseptic (Infections and infestations) | 6 | 2
Meningitis meningococcal (Infections and infestations) | 1 | 1
Meningitis pneumococcal (Infections and infestations) | 0 | 2
Meningitis viral (Infections and infestations) | 1 | 1
Myiasis (Infections and infestations) | 1 | 4
Nasal abscess (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 6 | 3
Necrotising fasciitis (Infections and infestations) | 0 | 1
Nosocomial infection (Infections and infestations) | 1 | 3
Oral candidiasis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 11 | 2
Osteomyelitis (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 4 | 8
Otitis media acute (Infections and infestations) | 16 | 16
Paronychia (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 12 | 16
Peritonitis (Infections and infestations) | 4 | 4
Pertussis (Infections and infestations) | 19 | 16
Pharyngeal abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 5 | 13
Pharyngotonsillitis (Infections and infestations) | 4 | 2
Pneumococcal sepsis (Infections and infestations) | 1 | 2
Pneumocystis jiroveci infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 478 | 557
Pneumonia adenoviral (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 2 | 5
Pneumonia viral (Infections and infestations) | 8 | 9
Postoperative wound infection (Infections and infestations) | 2 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 11 | 6
Pyelonephritis acute (Infections and infestations) | 2 | 1
Pyoderma (Infections and infestations) | 4 | 8
Pyomyositis (Infections and infestations) | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 6 | 5
Respiratory syncytial virus bronchitis (Infections and infestations) | 3 | 6
Respiratory syncytial virus infection (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 5 | 7
Roseola (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 1 | 0
Scarlet fever (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 11 | 14
Sepsis syndrome (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 4 | 7
Shigella infection (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 9 | 5
Skin candida (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 2 | 1
Staphylococcal scalded skin syndrome (Infections and infestations) | 3 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 1
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 2 | 0
Subcutaneous abscess (Infections and infestations) | 8 | 14
Systemic candida (Infections and infestations) | 2 | 1
Thyroglossal cyst infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 4 | 3
Tooth abscess (Infections and infestations) | 2 | 0
Tracheitis (Infections and infestations) | 8 | 7
Typhoid fever (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 15 | 11
Urinary tract infection (Infections and infestations) | 76 | 93
Urosepsis (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 10 | 18
Viral infection (Infections and infestations) | 12 | 11
Viral pharyngitis (Infections and infestations) | 9 | 7
Viral rash (Infections and infestations) | 3 | 4
Viral sepsis (Infections and infestations) | 0 | 1
Viral tonsillitis (Infections and infestations) | 0 | 1
Vulvovaginitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 3
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1
Accidental exposure (Injury, poisoning and procedural complications) | 10 | 8
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Accidental poisoning (Injury, poisoning and procedural complications) | 3 | 3
Animal bite (Injury, poisoning and procedural complications) | 5 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 6 | 5
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Burns first degree (Injury, poisoning and procedural complications) | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 6 | 8
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 2 | 1
Chemical injury (Injury, poisoning and procedural complications) | 1 | 0
Chemical poisoning (Injury, poisoning and procedural complications) | 24 | 21
Chest injury (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 39 | 36
Electric shock (Injury, poisoning and procedural complications) | 4 | 1
Electrical burn (Injury, poisoning and procedural complications) | 1 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Eye burns (Injury, poisoning and procedural complications) | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0
Eyelid injury (Injury, poisoning and procedural complications) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 5
Foreign body (Injury, poisoning and procedural complications) | 16 | 15
Fracture (Injury, poisoning and procedural complications) | 1 | 1
Gingival injury (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 2 | 3
Head injury (Injury, poisoning and procedural complications) | 75 | 74
Herbal toxicity (Injury, poisoning and procedural complications) | 2 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 4 | 2
Injury (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 2 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 2
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Mouth injury (Injury, poisoning and procedural complications) | 1 | 2
Multiple injuries (Injury, poisoning and procedural complications) | 26 | 33
Near drowning (Injury, poisoning and procedural complications) | 6 | 3
Open fracture (Injury, poisoning and procedural complications) | 0 | 2
Open wound (Injury, poisoning and procedural complications) | 1 | 0
Pneumonitis chemical (Injury, poisoning and procedural complications) | 1 | 3
Poisoning (Injury, poisoning and procedural complications) | 3 | 2
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2
Skull fracture (Injury, poisoning and procedural complications) | 6 | 5
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 25 | 36
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 2
Tongue injury (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 12 | 12
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 3 | 4
Vulvovaginal injury (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 5
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Acid base balance abnormal (Investigations) | 1 | 0
Aspiration bronchial (Investigations) | 2 | 3
Cow's milk intolerance (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 463 | 438
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 8 | 5
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Feeding disorder neonatal (Metabolism and nutrition disorders) | 0 | 1
Food intolerance (Metabolism and nutrition disorders) | 0 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 5
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 3 | 4
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Periostitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 3 | 2
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatoblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nephroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Retinoblastoma bilateral (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ataxia (Nervous system disorders) | 2 | 2
Brain injury (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Cerebrospinal fistula (Nervous system disorders) | 1 | 0
Cns ventriculitis (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 28 | 25
Dystonia (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 2 | 2
Extrapyramidal disorder (Nervous system disorders) | 2 | 0
Febrile convulsion (Nervous system disorders) | 95 | 135
Grand mal convulsion (Nervous system disorders) | 0 | 1
Guillain-barre syndrome (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Infantile spasms (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Myoclonic epilepsy (Nervous system disorders) | 0 | 1
Post-traumatic epilepsy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Viith nerve paralysis (Nervous system disorders) | 0 | 1
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Agitation (Psychiatric disorders) | 0 | 1
Binge eating (Psychiatric disorders) | 1 | 0
Breath holding (Psychiatric disorders) | 2 | 6
Psychomotor retardation (Psychiatric disorders) | 0 | 1
Glomerulonephritis acute (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 3 | 4
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 2 | 3
Oliguria (Renal and urinary disorders) | 1 | 0
Prerenal failure (Renal and urinary disorders) | 1 | 0
Pyelocaliectasis (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0
Genital lesion (Reproductive system and breast disorders) | 1 | 0
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 82 | 83
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 192 | 210
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 10 | 5
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 16 | 14
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 127 | 141
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Infantile asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 48 | 42
Acute haemorrhagic oedema of infancy (Skin and subcutaneous tissue disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 2 | 3
Cutaneous loxoscelism (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 2
Haemorrhagic urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 1
Henoch-schonlein purpura (Skin and subcutaneous tissue disorders) | 5 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rash scarlatiniform (Skin and subcutaneous tissue disorders) | 0 | 1
Skin oedema (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 10 | 15
Alcohol use (Social circumstances) | 0 | 1
Physical abuse (Social circumstances) | 1 | 2
Finger amputation (Surgical and medical procedures) | 1 | 0
Therapeutic hypothermia (Surgical and medical procedures) | 0 | 1
Toe amputation (Surgical and medical procedures) | 0 | 1
Capillary fragility (Vascular disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 3 | 3
Kawasaki's disease (Vascular disorders) | 9 | 3
Phlebitis (Vascular disorders) | 1 | 1
Shock (Vascular disorders) | 2 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Synflorix Group (N=3602) | Control Group (N=3612)
Anaemia (Blood and lymphatic system disorders) | 1411 | 1378
Conjunctivitis (Eye disorders) | 598 | 575
Diarrhoea (Gastrointestinal disorders) | 1905 | 1794
Vomiting (Gastrointestinal disorders) | 520 | 506
Constipation (Gastrointestinal disorders) | 279 | 257
Stomatitis (Gastrointestinal disorders) | 174 | 202
Injection site pain (General disorders) | 384 | 201
Pyrexia (General disorders) | 2272 | 1916
Irritability (General disorders) | 458 | 372
Injection site erythema (General disorders) | 260 | 172
Hypersensitivity (Immune system disorders) | 315 | 328
Nasopharyngitis (Infections and infestations) | 3338 | 3326
Gastroenteritis (Infections and infestations) | 1310 | 1281
Bronchiolitis (Infections and infestations) | 1119 | 1123
Pharyngitis (Infections and infestations) | 950 | 958
Viral infection (Infections and infestations) | 714 | 738
Pharyngotonsillitis (Infections and infestations) | 672 | 682
Rhinitis (Infections and infestations) | 542 | 516
Impetigo (Infections and infestations) | 497 | 474
Bronchitis (Infections and infestations) | 486 | 410
Pyoderma (Infections and infestations) | 350 | 368
Tonsillitis (Infections and infestations) | 232 | 232
Pneumonia (Infections and infestations) | 217 | 238
Urinary tract infection (Infections and infestations) | 202 | 228
Influenza (Infections and infestations) | 206 | 175
Head injury (Injury, poisoning and procedural complications) | 454 | 406
Malnutrition (Metabolism and nutrition disorders) | 556 | 545
Overweight (Metabolism and nutrition disorders) | 416 | 422
Dehydration (Metabolism and nutrition disorders) | 182 | 207
Asthma (Respiratory, thoracic and mediastinal disorders) | 596 | 582
Cough (Respiratory, thoracic and mediastinal disorders) | 499 | 510
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 288 | 313
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 322 | 297
Dermatitis (Skin and subcutaneous tissue disorders) | 468 | 464
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 293 | 316
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 332 | 296
Rash (Skin and subcutaneous tissue disorders) | 220 | 220
Prurigo (Skin and subcutaneous tissue disorders) | 179 | 199
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 163 | 196
Pain (General disorders) | 275/368 | 0/0 — AE collected in subjects in the Immunogenicity and Tolerability Subset post primary vaccination with Synflorix. Collect of results did not apply to subjects in the Control Group.
Pain (General disorders) | 270/368 | 0/0 — AE collected in subjects in the Immunogenicity and Tolerability Subset post primary vaccination with Infanrix Hexa. Collect of results did not apply to subjects in the Control Group.
Redness (General disorders) | 182/368 | 0/0 — AE collected in subjects in the Immunogenicity and Tolerability Subset post primary vaccination with Synflorix. Collect of results did not apply to subjects in the Control Group.
Redness (General disorders) | 171/368 | 0/0 — AE collected in subjects in the Immunogenicity and Tolerability Subset post primary vaccination with Infanrix Hexa. Collect of results did not apply to subjects in the Control Group.
Redness (General disorders) | 0/0 | 118/357 — AE collected in subjects in the Immunogenicity and Tolerability Subset post primary vaccination with Infanrix-IPV/Hib. Collect of results did not apply to subjects in the Synflorix Group.
Redness (General disorders) | 0/0 | 109/357 — AE collected in subjects in the Immunogenicity and Tolerability Subset post primary vaccination with Engerix. Collect of results did not apply to subjects in the Synflorix Group.
Swelling (General disorders) | 141/368 | 0/0 — AE collected in subjects in the Immunogenicity and Tolerability Subset post primary vaccination with Synflorix. Collect of results did not apply to subjects in the Control Group.
Swelling (General disorders) | 143/368 | 0/0 — AE collected in subjects in the Immunogenicity and Tolerability Subset post primary vaccination with Infanrix Hexa. Collect of results did not apply to subjects in the Control Group.
Swelling (General disorders) | 0/0 | 98/357 — AE collected in subjects in the Immunogenicity and Tolerability Subset post primary vaccination with Infanrix-IPV/Hib. Collect of results did not apply to subjects in the Synflorix Group.
Swelling (General disorders) | 0/0 | 91/357 — AE collected in subjects in the Immunogenicity and Tolerability Subset post primary vaccination with Engerix. Collect of results did not apply to subjects in the Synflorix Group.
Pain (General disorders) | 129/317 | 0/0 — AE collected in subjects in the Immunogenicity and Tolerability Subset post booster vaccination with Synflorix. Collect of results did not apply to subjects in the Control Group.
Pain (General disorders) | 317/317 | 81/303 — AE collected in subjects in the Immunogenicity and Tolerability Subset post booster vaccination with Infanrix-IPV/Hib.
Pain (General disorders) | 0/0 | 89/303 — AE collected in subjects in the Immunogenicity and Tolerability Subset post booster vaccination with Havrix. Collect of results did not apply to subjects in the Synflorix Group.
Redness (General disorders) | 104/317 | 0/0 — AE collected in subjects in the Immunogenicity and Tolerability Subset post booster vaccination with Synflorix. Collect of results did not apply to subjects in the Control Group.
Redness (General disorders) | 98/317 | 81/303 — AE collected in subjects in the Immunogenicity and Tolerability Subset post booster vaccination with Infanrix-IPV/Hib.
Redness (General disorders) | 0/0 | 73/303 — AE collected in subjects in the Immunogenicity and Tolerability Subset post booster vaccination with Havrix. Collect of results did not apply to subjects in the Synflorix Group.
Swelling (General disorders) | 74/317 | 0/0 — AE collected in subjects in the Immunogenicity and Tolerability Subset post booster vaccination with Synflorix. Collect of results did not apply to subjects in the Control Group.
Swelling† (General disorders) | 69/317 | 70/303 — AE collected in subjects in the Immunogenicity and Tolerability Subset post booster vaccination with Infanrix-IPV/Hib.
Swelling (General disorders) | 0/0 | 55/303 — AE collected in subjects in the Immunogenicity and Tolerability Subset post booster vaccination with Havrix. Collect of results did not apply to subjects in the Synflorix Group.
Drowsiness (General disorders) | 236/368 | 168/357 — AE collected in subjects in the Immunogenicity and Tolerability Subset post primary vaccination
Fever (rectal temperature >= 38.0°C) (General disorders) | 247/368 | 125/357 — AE collected in subjects in the Immunogenicity and Tolerability Subset post primary vaccination
Irritability (General disorders) | 289/368 | 206/357 — AE collected in subjects in the Immunogenicity and Tolerability Subset post primary vaccination
Loss of appetite (General disorders) | 133/368 | 80/357 — AE collected in subjects in the Immunogenicity and Tolerability Subset post primary vaccination
Drowsiness (General disorders) | 74/317 | 65/303 — AE collected in subjects in the Immunogenicity and Tolerability Subset post booster vaccination
Fever (rectal temperature >= 38.0°C) (General disorders) | 93/317 | 73/303 — AE collected in subjects in the Immunogenicity and Tolerability Subset post booster vaccination
Irritability (General disorders) | 121/317 | 95/303 — AE collected in subjects in the Immunogenicity and Tolerability Subset post booster vaccination
Loss of appetite (General disorders) | 51/317 | 46/303 — AE collected in subjects in the Immunogenicity and Tolerability Subset post booster vaccination
PAIN (General disorders) | 0/0 | 169/357 — AE collected in subjects in the Immunogenicity and Tolerability Subset post primary vaccination with Infanrix-IPV/Hib. Collect of results did not apply to subjects in the Synflorix Group.
PAIN (General disorders) | 0/0 | 165/357 — AE collected in subjects in the Immunogenicity and Tolerability Subset post primary vaccination with Engerix. Collect of results did not apply to subjects in the Synflorix Group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.